CLINICAL TRIAL: NCT01797835
Title: Alcohol Screening in an Ethnically Diverse Sample of Adolescents in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Valley Community Clinic (Unknown); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01AA021786 (NIH)
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Use; Drug Use
Keywords: adolescents; intervention; motivational interviewing; alcohol and drug use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Placebo Comparator): Youth in usual care will receive screening for alcohol and drug use. Those youth who are at risk will have a chance to talk to their provider about their use. They will also receive an informational brochure.
  Interventions: Behavioral: usual care
- CHAT brief MI intervention (Experimental): Youth in CHAT will receive screening for alcohol and drug use. Those youth who are at risk will have a chance to talk to their provider about their use. In addition, these youth will CHAT. CHAT is a brief motivational intervention that takes places in the primary care setting. It is a 15-20 minute intervention for adolescents age 12-18 focused on discussing alcohol and drug use. They will also receive a booster call one month later to check in on how they are doing.
  Interventions: Behavioral: CHAT brief MI intervention

INTERVENTIONS:
Behavioral: CHAT brief MI intervention — CHAT is one 15-20 minute session delivered in a single PC visit and utilizes motivational interviewing with youth to target alcohol and drug use in primary care.
  Arms: CHAT brief MI intervention
Behavioral: usual care — Youth receive a brochure with information on AOD use.
  Arms: Usual Care

SUMMARY:
Screening youth in the primary care setting is one way to identify adolescents who may be at-risk for future alcohol problems. The current study tests the new NIAAA screening guide questions, which ask about friend and adolescent drinking, to see how well these questions work to predict subsequent alcohol use, problems, and involvement in other risk behaviors, such as sexual risk-taking and delinquency. In addition, the investigators plan to provide a brief motivational intervention for some at-risk teens and see whether alcohol use differs for those teens who receive the intervention and those teens who receive enhanced usual care. The results of this study have the potential to significantly impact the standard of care for identifying and intervening with at- risk youth in primary care settings.

ELIGIBILITY:
Inclusion Criteria: 1

* 12-18
* speak English

Exclusion Criteria:

* cognitive impairment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 294 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J D'Amico, PhD, Principal Investigator — RAND
Locations (2):
- United States (2):
  - Valley Community Clinic, North Hollywood, California
  - UPMC St. Margaret, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] D'Amico EJ, Parast L, Osilla KC, Seelam R, Meredith LS, Shadel WG, Stein BD. Understanding Which Teenagers Benefit Most From a Brief Primary Care Substance Use Intervention. Pediatrics. 2019 Aug;144(2):e20183014. doi: 10.1542/peds.2018-3014. Epub 2019 Jul 11. PMID 31296568
- [Derived] Meredith LS, Seelam R, Stein BD, Parast L, Shadel WG, D'Amico EJ. Adolescents with better mental health have less problem alcohol use six months later. Addict Behav. 2019 Aug;95:77-81. doi: 10.1016/j.addbeh.2019.03.006. Epub 2019 Mar 7. PMID 30861475
- [Derived] D'Amico EJ, Parast L, Shadel WG, Meredith LS, Seelam R, Stein BD. Brief motivational interviewing intervention to reduce alcohol and marijuana use for at-risk adolescents in primary care. J Consult Clin Psychol. 2018 Sep;86(9):775-786. doi: 10.1037/ccp0000332. PMID 30138016
- [Derived] Meredith LS, Ewing BA, Stein BD, Shadel WG, Brooks Holliday S, Parast L, D'Amico EJ. Influence of mental health and alcohol or other drug use risk on adolescent reported care received in primary care settings. BMC Fam Pract. 2018 Jan 9;19(1):10. doi: 10.1186/s12875-017-0689-y. PMID 29316897
- [Derived] D'Amico EJ, Parast L, Meredith LS, Ewing BA, Shadel WG, Stein BD. Screening in Primary Care: What Is the Best Way to Identify At-Risk Youth for Substance Use? Pediatrics. 2016 Dec;138(6):e20161717. doi: 10.1542/peds.2016-1717. Epub 2016 Nov 18. PMID 27940696

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: this study included an examination of screening; thus, not all youth were part of the randomized controlled trial as they screened in at low risk. This is why there is a larger N for the overall sample. The 294 are the youth that screened in as at-risk who were then part of the RCT.
Period: Overall Study
Arm/Group | CHAT Brief MI Intervention | Usual Care
Started | 153 | 141
Completed | 122 | 114
Not Completed | 31 | 27
Not completed — Lost to Follow-up | 31 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHAT Brief MI Intervention | Usual Care | Total
Number analyzed (Participants) | 153 | 141 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] — asked how old they were
  years | 16.16 (1.61) | 15.91 (1.61) | 16 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 77 | 167
  Male | 63 | 64 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 96 | 195
  Not Hispanic or Latino | 54 | 45 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 18 | 49
  White | 118 | 111 | 229
  More than one race | 4 | 12 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 153 | 141 | 294

OUTCOME MEASURES:

1. Primary Outcome: Number of Times Used Alcohol
Description: in the past three months: Number of times used alcohol; The 6-point frequency response scale (0= "Never" to 5= "More than 20 times") was rescaled to a pseudo-continuous variable ranging from 0 to 20 using the mid-point of any range as the new value (e.g. 3-10 times was recoded as 6.5 times).
Time Frame: Past 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Care | CHAT Brief MI Intervention
Number analyzed (Participants) | 141 | 153
score on a scale | 5.64 [0 to 20] | 5.18 [0 to 20]

2. Secondary Outcome: Number of Times Used Marijuana
Description: number of times used marijuana in the past 3 months; The 6-point frequency response scale (0= "Never" to 5= "More than 20 times") was rescaled to a pseudo-continuous variable ranging from 0 to 20 using the mid-point of any range as the new value (e.g. 3-10 times was recoded as 6.5 times).
Time Frame: Past 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Care | CHAT Brief MI Intervention
Number analyzed (Participants) | 141 | 153
score on a scale | 5.95 [0 to 20] | 6.38 [0 to 20]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Event (AE): any untoward medical occurrence that may present itself during treatment or administration of an intervention, and which may or may not have a causal relationship with the treatment. Adverse events could arise from the study (e.g., breach of confidentiality) or could arise due to the population under study (e.g., a youth reports extensive use of drugs or that he/she "huffs" daily).
Arm/Group | Usual Care | CHAT Brief MI Intervention
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/153
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/153
Other Adverse Events (participants affected / at risk) | 0/141 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT01797835/Prot_SAP_000.pdf